CLINICAL TRIAL: NCT02041910
Title: Testicular Injection of Autologous Human Bone Marrow Derived Stem Cells for Treatment of Patients With Azoospermia
Brief Title: Testicular Injection of Autologous Stem Cells for Treatment of Patients With Azoospermia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hesham Saeed Elshaer (Other)
Responsible Party: Sponsor-Investigator, Hesham Saeed Elshaer, Associate Professor & Director, El-Rayadh Fertility Centre
Organization: El-Rayadh Fertility Centre (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCT0550330; RFC0550330 (Other Grant/Funding Number: RayadhFC0550330)
Record Dates: First submitted 2014-01-10; First posted 2014-01-22 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Azoospermia
MeSH Terms: conditions — Azoospermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stem Cells (Experimental): 60 ml of Bone marrow will aspirated for stem cells isolation and preparation. 5 ml of stem cells prepared according to GMP rules injected into testis.
  Interventions: Biological: Stem Cells
- Stem Cells Injection (Experimental): Stem Cell Dose 3-5 Million Autologous MSCs Injected into testis.
  Interventions: Biological: Stem Cells

INTERVENTIONS:
Biological: Stem Cells — MSCs injection intratesticular
  Other Names: MSCs
  Arms: Stem Cells
Biological: Stem Cells — 60 ml of Bone marrow will aspirated for stem cells isolation and preparation. 5 ml of stem cells prepared according to GMP rules injected into testis.
  Arms: Stem Cells Injection

SUMMARY:
Azoospermia is defined as the complete lack of sperm in the ejaculate. In humans, Azoospermia affects about 1% of the male population and may be seen in up to 20% of male infertility situations. In testicular Azoospermia the testes are abnormal, atrophic, or absent, and sperm production severely disturbed to absent. FSH levels tend to be elevated (hypergonadotropic) as the feedback loop is interrupted. The condition is seen in 49-93% of men with Azoospermia. The purpose of this study is to assess the ability of bone marrow derived stem cells to differentiate into germ cells and their role in treatment of testicular Azoospermia

DETAILED DESCRIPTION:
This study is an open-label investigation of the efficacy of injection autologous adult bone marrow derived stem cells into the somniferous tubules or interstitial spaces of male testis with Azospermia. Sixty men with Azoospermia will be recruited in this study after a written informed consent.

The diagnosis of Azoospermia will be established on the basis of two semen analysis evaluations done at separate occasions; this will be followed by detailed history taking, physical examination and investigations. History taking will include general health, sexual health, past fertility, libido, sexual activity and previous exposure to surgery, drugs, mumps infection and irradiation. Physical examination includes genital and local examination for detection of signs of Klinefelter syndrome, testicular atrophy, absence of vas. Investigations include serum FSH, LH, karyotyping and testosterone levels, and may include testicular biopsy or transrectal ultrasound if indicated (Low levels of LH and FSH with low or normal testosterone levels are indicative of pretesticular problems, while high levels of gonadotropins indicate testicular problems. However, often this distinction is not clear and the differentiation between obstructive versus non-obstructive Azoospermia may require a testicular biopsy).

Subjects will be enrolled based on specific inclusion/exclusion criteria and evaluated at regular post transplant intervals. Human adult bone marrow derived stem cells will be transplanted by an andrological surgeon through a standard surgical approach. Subjects will be monitored frequently for a total of one year after adult bone marrow stem cells cell injection. For safety of participants, Bone Marrow Stem cells will be injected in one testis only and the other testis will be spared.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-obstructive Azoospermia
* Patients between 25 - 60 years old.

Exclusion Criteria:

* Patients with obstructive Azoospermia
* Men with previous surgery in testis
* Men with infectious genital diseases and anatomical abnormalities of the genital tract
* Those with major medical problems such as malignancy, hepatitis, etc.
* Chromosomal aberration (e.g. Y microdeleion, trisomy….)

Ages: 25 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Cases Improvement | 12 Weeks
  Serum Hormonal Profile:
  (elevation of testosterone levels, decreasing of FSH, LH and Prolactine Levels); Testicular Size (increased size); and Sexual Potency (increased sexual potency).

SECONDARY OUTCOMES:
Cases Improvement | 48 Weeks
  Testicular biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Taimour Khalifa, MD, Principal Investigator — Al-Azhar University; Sayed Bakry, PhD, Study Director — Al-Azhar University; Hala Gabr, MD, Study Chair — Cairo University; Wael Abu El Khier, MD, Study Chair — Military Academy
Locations (1):
- El-Rayadh Fertility Center, Al Mohandseen, Giza Governorate, Egypt